CLINICAL TRIAL: NCT03372369
Title: A Randomized Control Trial of the Effectiveness of Risk Communication in Two Contraceptive Fact Sheets
Brief Title: Testing the Impact of Two Posters on Contraceptive Knowledge, Contraceptive Preferences, and Perceived Pregnancy Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-2955; UL1TR001111 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-13 (Actual); Results first posted 2019-06-07 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2017-12

CONDITIONS: Contraception; Knowledge, Attitudes, Practice
Keywords: contraceptive knowledge; contraceptive use; educational intervention; poster; online survey
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDC Poster (Active Comparator): After collecting baseline contraceptive knowledge, method preference, if participant were to switch methods during the next year, and current perceived pregnancy risk, participants will view CDC poster for contraceptive effectiveness.
  Interventions: Other: View CDC Poster
- Patient-Centered Poster (Experimental): After collecting baseline contraceptive knowledge, method preference, if participant were to switch methods during the next year, and current perceived pregnancy risk, participants will view Patient-Centered poster for contraceptive effectiveness.
  Interventions: Other: View Patient-Centered Poster

INTERVENTIONS:
Other: View CDC Poster — The poster designed by the CDC to explain contraceptive effectiveness.
  Arms: CDC Poster
Other: View Patient-Centered Poster — The poster designed by the research team to explain contraceptive effectiveness. This poster was developed through cognitive interviews with 26 North Carolina women, and the final version of this poster was found to be more useful, acceptable, and attractive than the CDC poster by the majority of women participating.
  Arms: Patient-Centered Poster

SUMMARY:
This study tests two posters that teach people about contraception: one designed by the Centers for Disease Control (CDC), and one designed by the researchers. The investigators hypothesize that the new poster will have more increased (1) contraceptive knowledge, (2) willingness to use effective contraception, and (3) perceived pregnancy risk than the CDC poster. This study will expand useful knowledge because contraceptive knowledge, willingness to use effective contraception, and perceived pregnancy risk have been shown to affect women's likelihood of using contraception. If the investigators learn how to increase these factors, the investigators could theoretically reduce women's risk of unplanned pregnancy.

The investigators will test this hypothesis by recruiting N=1000 women to complete an online survey using Amazon Mechanical Turk. These women will complete a survey that will first measure their initial contraceptive knowledge, willingness to use effective contraception, and perceived pregnancy risk. Then women will randomly be shown one of the two posters. Then, the investigators will measure their contraceptive knowledge, willingness to use effective contraception, and perceived pregnancy risk again. The investigators will use statistical tests (a t-test) to find out whether there are significant changes in these three outcomes for either of the posters, and whether one poster does a better job of changing these outcomes than the other.

DETAILED DESCRIPTION:
Purpose: To evaluate the effectiveness of two posters' ability to improve contraceptive knowledge, willingness to use effective contraception, and pregnancy risk perceptions. One of these posters was developed by the CDC. The other was developed by the research team in a previous study using cognitive interviews with N=26 women. The new poster is designed to meet the informational needs of women with low numeracy (i.e. low facility with math) and women who do not use contraception.

Participants: The investigators will recruit N=1020 women aged 18-44 who can speak and read English, have been sexually active in the last three months, and who are not pregnant or trying to get pregnant.

Procedures (methods): The investigators will use Amazon Mechanical Turk to recruit participants. Participants will take one survey. The survey will first ask baseline questions to assess contraceptive knowledge, willingness to use effective contraception, and perceived pregnancy risk. Participants will then be randomly shown one of the two posters. Then post-exposure questions on the three outcomes will be asked.

The investigators test the hypotheses that before compared to after exposure, the mean scores for (1) contraceptive knowledge, (2) willingness to use effective contraception, and (3) perceived pregnancy risk will increase more for the new fact sheet than for the CDC sheet.

The investigators also collect the following covariates: age, race/ethnicity, education, income, insurance type, insurance coverage of contraception, numeracy (facility with math), health and safety contraindications to contraceptive use, sexual orientation, parenthood, years since first sex, relationship status, prior exposure to CDC sheet, and pregnancy avoidance intensity. The investigators will compare whether the covariates are balanced between the randomized groups and the US population using two-sample t-tests, chi-squared, or nonparametric tests as appropriate. If the unbalance is statistically significant, the investigators will include the covariate in the regression to compare the adjusted difference between treatments. The investigators use two-sample t-tests to test our hypotheses. The investigators will also test for subgroup differences in our outcomes based on our covariates using a Chow test.

The investigators will first test survey mechanics (correct coding, correct links) on N=20 women. The investigators will survey N=1000 women for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Speak and read English
* Have had vaginal intercourse in the past three months

Exclusion Criteria:

* Are pregnant
* Are trying to conceive

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 990 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seri AL Anderson, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Kristen H Lich, PHD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of individual participant data with other researchers

REFERENCES:
- [Derived] Anderson S, Frerichs L, Kaysin A, Wheeler SB, Halpern CT, Lich KH. Effects of Two Educational Posters on Contraceptive Knowledge and Intentions: A Randomized Controlled Trial. Obstet Gynecol. 2019 Jan;133(1):53-62. doi: 10.1097/AOG.0000000000003012. PMID 30531560

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between January 26 and February 13, 2018. They were enrolled and participated in the study through a survey distributed on Amazon Mechanical Turk.
Period: Qualification Period
Arm/Group | CDC Poster | Patient-Centered Poster
Started | 495 | 495
Completed | 469 | 473
Not Completed | 26 | 22
Not completed — Withdrawal by Subject | 16 | 13
Not completed — Inconsistent Eligibility Results | 10 | 9
Period: Intervention and Follow-Up Period
Arm/Group | CDC Poster | Patient-Centered Poster
Started | 469 | 473
Completed | 466 | 470
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Population: Baseline data is reported for participants completing the qualification phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | CDC Poster | Patient-Centered Poster | Total
Number analyzed (Participants) | 469 | 473 | 942
Age, Continuous [Mean (Full Range); unit: years] | 32 [18 to 44] | 32 [18 to 44] | 32 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 469 | 473 | 942
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnicity: White | 353 | 351 | 704
  Race or Ethnicity: Black or African American | 45 | 36 | 81
  Race or Ethnicity: Hispanic or Latina | 17 | 21 | 38
  Race or Ethnicity: Some Other Race | 28 | 34 | 62
  Race or Ethnicity: Multiracial | 26 | 31 | 57
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 469 | 473 | 942

OUTCOME MEASURES:

1. Primary Outcome: Change in Contraceptive Knowledge Assessment (CKA) Score
Description: The CKA is a 25-item tool covering knowledge gaps like long-acting reversible contraceptives, emergency contraception, common myths, and efficacy rates which will be used to determine contraception knowledge. One point is added for each correctly answered question for a total possible score of 25. Higher scores reflect greater contraceptive knowledge.
Time Frame: Baseline and 15-20 minutes after baseline (3 minutes after exposure to a poster)
Measure: Mean (99% Confidence Interval); unit: scores on a scale
Arm/Group | CDC Poster | Patient-Centered Poster
Number analyzed (Participants) | 466 | 470
scores on a scale | 0.90 [0.66 to 1.13] | 1.6 [1.31 to 1.90]
Statistical Analysis 1: Comparison: CDC Poster; The null hypothesis is that the change in the contraceptive knowledge score for the CDC poster between baseline and followup is 0; Test type: Superiority; p < 0.0001, t-test, 1 sided — The Bonferroni correction is used to account for multiple comparisons. In this analysis, p<0.01 is the threshold for statistical significance
Statistical Analysis 2: Comparison: Patient-Centered Poster; The null hypothesis is that the change in the contraceptive knowledge score for the patient-centered poster between baseline and followup is 0; Test type: Superiority; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: CDC Poster vs Patient-Centered Poster; The null hypothesis is that the patient-centered poster does not produce a larger increase in the contraceptive knowledge score between baseline and followup than the CDC poster; Test type: Superiority; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Change in Effective Contraception Preference Score
Description: Women will be asked whether they are planning on switching contraceptive methods in the next year and which methods of contraception they would hypothetically consider using if they were to switch contraceptive methods within the next year. They are then asked to rank the methods in order of how likely they would be to use each method. A woman's "contraceptive preference" is the method that she says she would be most likely to use. Methods will be scored from 0-3: '0' for no method, '1' for ineffective methods like condoms, '2' for effective methods like the Pill, and '3' for highly effective methods like Intrauterine Devices (IUDs). Positive scores reflect improvements in the effectiveness of the contraceptive method that women say they are likely to use.
Time Frame: Baseline and 15-20 minutes after baseline (1 minute after exposure to a poster)
Measure: Mean (99% Confidence Interval); unit: scores on a scale
Arm/Group | CDC Poster | Patient-Centered Poster
Number analyzed (Participants) | 466 | 470
scores on a scale | 0.09 [0.02 to 0.17] | 0.09 [0.01 to 0.17]
Statistical Analysis 1: Comparison: CDC Poster; The null hypothesis is that the change in the effective contraception preference score for the CDC poster between baseline and followup is 0; Test type: Superiority; p < 0.001, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Patient-Centered Poster; The null hypothesis is that the change in the effective contraception preference score for the patient-centered poster between baseline and followup is 0; Test type: Superiority; p < 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: CDC Poster vs Patient-Centered Poster; The null hypothesis is that the patient-centered poster does not produce a larger increase in the effective contraception preference score between baseline and followup than the CDC poster; Test type: Superiority; p > 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]

3. Primary Outcome: Change in Perceived Pregnancy Risk Score
Description: Women are asked what their chances of getting pregnant this year are (very high=4, high=3, moderate=2, low=1, very low=0). A good outcome in terms of reducing the risk of unprotected sex and unplanned pregnancy would be increased perceived pregnancy risk as reflected in a higher score.
Time Frame: Baseline and 15-20 minutes after baseline (2 minutes after exposure to a poster)
Measure: Mean (99% Confidence Interval); unit: scores on a scale
Arm/Group | CDC Poster | Patient-Centered Poster
Number analyzed (Participants) | 466 | 470
scores on a scale | 0.002 [-0.06 to 0.06] | 0.03 [-0.03 to 0.09]
Statistical Analysis 1: Comparison: CDC Poster; The null hypothesis is that the change in the perceived pregnancy risk score for the CDC poster between baseline and followup is 0; Test type: Superiority; p > 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Patient-Centered Poster; The null hypothesis is that the change in the perceived pregnancy risk score for the patient-centered poster between baseline and followup is 0; Test type: Superiority; p > 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: CDC Poster vs Patient-Centered Poster; The null hypothesis is that the patient-centered poster does not produce a larger increase in the perceived pregnancy risk score between baseline and followup than the CDC poster; Test type: Superiority; p > 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]

4. Post Hoc Outcome: Change in Mean Accuracy of Perceived Pregnancy Risk Score
Description: Women are asked what their chances of getting pregnant this year are (very high, high, moderate, low, very low). This response is compared to the most effective contraceptive method women reported using in the past three months using the same categories of effectiveness as in the "change in effective contraception preference score" outcome. Women received a score of 1 if their perceived pregnancy risk was accurate based on their current contraceptive method and a score of 0 if it was inaccurate. Women's perceived pregnancy risk was accurate if: they used a highly effective method and they said they were at very low risk; if they used an effective method and they said they were at low or moderate risk; if they used a less effective method and said they were at moderate or high risk; or if they used no method and said they were at very high risk. A good outcome would be increased accuracy of perceived pregnancy risk as reflected by a higher score.
Time Frame: Baseline and 15-20 minutes after baseline (2 minutes after exposure to a poster)
Measure: Mean (99% Confidence Interval); unit: scores on a scale
Arm/Group | CDC Poster | Patient-Centered Poster
Number analyzed (Participants) | 466 | 470
scores on a scale | 0 [-0.02 to 0.02] | 0.013 [-0.01 to 0.04]
Statistical Analysis 1: Comparison: CDC Poster; The null hypothesis is that the change in the accuracy of perceived pregnancy risk score for the CDC poster between baseline and followup is 0; Test type: Superiority; p > 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Patient-Centered Poster; The null hypothesis is that the change in the accuracy of perceived pregnancy risk score for the patient-centered poster between baseline and followup is 0; Test type: Superiority; p > 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: CDC Poster vs Patient-Centered Poster; The null hypothesis is that the patient-centered poster does not produce a larger increase in the accuracy of perceived pregnancy risk score between baseline and followup than the CDC poster; Test type: Superiority; p > 0.01, t-test, 1 sided — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Participants could report adverse events from the time they began the study survey through survey completion; up to 2 hours.
Description: No difference
Arm/Group | CDC Poster | Patient-Centered Poster
All-Cause Mortality (participants affected / at risk) | 0/495 | 0/495
Serious Adverse Events (participants affected / at risk) | 0/495 | 0/495
Other Adverse Events (participants affected / at risk) | 0/495 | 0/495

LIMITATIONS AND CAVEATS:
Results are likely only generalizable to US female internet users. The study does not assess the impact of the posters on behavior, only intentions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03372369/Prot_SAP_000.pdf